CLINICAL TRIAL: NCT03879928
Title: A Randomized, Double-blind, Placebo-controlled, Alternating Panel Single Ascending Dose, Sequential Multiple Ascending Dose, and Food Effect Study of FM101 in Healthy Male and Female Volunteers
Brief Title: A SAD, MAD, and FE Study to Evaluate the Safety, Tolerability, and Pharmacokinetic Profile of FM101 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Future Medicine (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: FM101-CTP1-001
Record Dates: First submitted 2019-03-12; First posted 2019-03-19 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (13):
- Placebo for SAD (Placebo Comparator): Placebo comparator for SAD
  Interventions: Drug: Single ascending doses of FM101
- FM101 75 mg for SAD (Experimental): Single ascending doses of FM101
  Interventions: Drug: Single ascending doses of FM101
- FM101 150 mg for SAD (Experimental): Single ascending doses of FM101
  Interventions: Drug: Single ascending doses of FM101
- FM101 300 mg for SAD (Experimental): Single ascending doses of FM101
  Interventions: Drug: Single ascending doses of FM101
- FM101 600 mg for SAD (Experimental): Single ascending doses of FM101
  Interventions: Drug: Single ascending doses of FM101
- FM101 1200 mg for SAD (Experimental): Single ascending doses of FM101
  Interventions: Drug: Single ascending doses of FM101
- FM101 2400 mg for SAD (Experimental): Single ascending doses of FM101
  Interventions: Drug: Single ascending doses of FM101
- Placebo for MAD (Placebo Comparator): Placebo comparator for MAD
  Interventions: Drug: Multiple ascending doses of FM101
- FM101 150 mg (QD) for MAD (Experimental): Multiple ascending doses of FM101
  Interventions: Drug: Multiple ascending doses of FM101
- FM101 450 mg (QD) for MAD (Experimental): Multiple ascending doses of FM101
  Interventions: Drug: Multiple ascending doses of FM101
- FM101 600 mg (BID) for MAD (Experimental): Multiple ascending doses of FM101
  Interventions: Drug: Multiple ascending doses of FM101
- FM101 300 mg under fasted condition for FE (Experimental): Food Effect of FM101
  Interventions: Drug: Food effects of FM101
- FM101 300 mg under fed condition for FE (Experimental): Food Effect of FM101
  Interventions: Drug: Food effects of FM101

INTERVENTIONS:
Drug: Single ascending doses of FM101 — The study drug (FM101 and placebo comparator) will be administered orally as SAD doses
  Arms: FM101 1200 mg for SAD; FM101 150 mg for SAD; FM101 2400 mg for SAD; FM101 300 mg for SAD; FM101 600 mg for SAD; FM101 75 mg for SAD; Placebo for SAD
Drug: Multiple ascending doses of FM101 — The study drug (FM101 and placebo comparator) will be administered orally as MAD doses
  Arms: FM101 150 mg (QD) for MAD; FM101 450 mg (QD) for MAD; FM101 600 mg (BID) for MAD; Placebo for MAD
Drug: Food effects of FM101 — The study drug (FM101) will be administered orally under fasted condition and fed condition.
  Arms: FM101 300 mg under fasted condition for FE; FM101 300 mg under fed condition for FE

SUMMARY:
This a double blind, randomized, placebo controlled, single and multiple ascending dose (SAD/MAD) study in healthy subjects. Safety evaluation will include adverse events (TEAEs), clinical laboratory values, vital signs, ECGs, and physical examinations.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study in healthy volunteers designed to assess the safety, tolerability and PK of FM101. This study will consist of 3 parts: a SAD part, a single dose FE part and a MAD part. Each subject is to participate in only 1 part of the study.

ELIGIBILITY:
Inclusion Criteria:

* Gender: male or female
* Age: 18 - 50 years, inclusive, at screening
* Body mass index (BMI) : 18.0 - 32.0 kg/m2 (inclusive)
* Weight : ≥ 50 kg
* Status : healthy subjects
* At screening, females must be non-pregnant and non-lactating, or of non child-bearing potential (either surgically sterilized or physiologically incapable of becoming pregnant, or at least 1 year post menopausal [amenorrhea duration of 12 consecutive months); non-pregnancy will be confirmed for all females by a serum pregnancy test conducted at screening, and a urine pregnancy test at each admission and at follow-up.
* Female subjects of child-bearing potential, with a fertile male sexual partner, must agree to use adequate contraception from screening until 90 days after the follow up visit. Adequate contraception is defined as using hormonal contraceptives or an intrauterine device combined with at least 1 of the following forms of contraception: a diaphragm or cervical cap, or a condom. Also, total abstinence, in accordance with the lifestyle of the subject, is acceptable.
* Male subjects, if not surgically sterilized, must agree to use adequate contraception and not donate sperm from first admission to the clinical research center until 90 days after the follow-up visit. Adequate contraception for the male subject (and his female partner) is defined as using hormonal contraceptives or an intrauterine device combined with at least 1 of the following forms of contraception: a diaphragm or cervical cap, or a condom. Also, total abstinence, in accordance with the lifestyle of the subject is acceptable.
* All prescribed medication must have been stopped at least 14 days prior to (each) admission to the clinical research center. An exception is made for hormonal contraceptives, which may be used throughout the study.
* All over-the-counter medication, vitamin preparations and other food supplements, or herbal medications (eg, St. John's Wort) must have been stopped at least 7 days prior to (each) admission to the clinical research center. An exception is made for paracetamol, which is allowed up to admission to the clinical research center.
* Ability and willingness to abstain from alcohol, methylxanthine-containing beverages or food (coffee, tea, cola, chocolate, energy drinks), grapefruit (juice), and tobacco products from 48 hours prior to (each) admission to the clinical research center.
* Good physical and mental health on the basis of medical history, physical examination, clinical laboratory, ECG, and vital signs, as judged by the Investigator.
* Willing and able to sign the ICF.

Exclusion Criteria:

* Employee of CRO or the Sponsor.
* History of relevant drug and/or food allergies.
* Using tobacco products within 60 days prior to (the first) drug administration.
* History of alcohol abuse or drug addiction (including soft drugs like cannabis products).
* Positive drug and alcohol screen (opiates, methadone, cocaine, amphetamines [including ecstasy], cannabinoids, barbiturates, benzodiazepines, gamma hydroxybutyric acid [GHB], tricyclic antidepressants, and alcohol) at screening and (each) admission to the clinical research center.
* Average intake of more than 24 units of alcohol per week (1 unit of alcohol equals approximately 250 mL of beer, 100 mL of wine, or 35 mL of spirits).
* Positive screen for hepatitis B surface antigen (HBsAg), anti hepatitis C virus (HCV) antibodies, or anti human immunodeficiency virus (HIV) 1 and 2 antibodies.
* Participation in a drug study within 60 days prior to (the first) drug administration in the current study. Participation in more than 3 other drug studies (for male subjects) / more than 2 other drug studies (for female subjects) in the 10 months prior to (the first) drug administration in the current study.
* Donation or loss of more than 100 mL of blood within 60 days prior to (the first) drug administration. Donation or loss of more than 1.5 liters of blood (for male subjects) / more than 1.0 liters of blood (for female subjects) in the 10 months prior to (the first) drug administration in the current study.
* Significant and/or acute illness within 5 days prior to (the first) drug administration that may impact safety assessments, in the opinion of the Investigator.
* Non-willingness to consume the high-fat breakfast (Part B only).
* Unsuitable veins for infusion or blood sampling.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2019-08-18 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of FM101 after SAD and MAD doses to healthy volunteers by assessing the number, severity, and type of TEAEs. | SAD [Day 1 through Day 7], MAD [Day 1 through Day 10]
  The number of TEAEs (frequency of occurrence, number of subjects experiencing the event)
To evaluate the change in clinical laboratory values from the baseline after SAD and MAD doses. | SAD [Day 1 through Day 7], MAD [Day 1 through Day 10]
  The number of abnormalities with clinical significance (frequency of occurrence, number of subjects experiencing the event)
To evaluate the change in vital signs from the baseline after SAD and MAD doses. | SAD [Day 1 through Day 7], MAD [Day 1 through Day 10]
  The number of abnormalities with clinical significance (frequency of occurrence, number of subjects experiencing the event)
To evaluate the change in electrocardiograms (ECGs) after SAD and MAD doses. | SAD [Day 1 through Day 7], MAD [Day 1 through Day 10]
  The number of abnormalities with clinical significance (frequency of occurrence, number of subjects experiencing the event).
To evaluate the change in physical examinations after SAD and MAD doses. | SAD [Day 1 through Day 7], MAD [Day 1 through Day 10]
  The number of abnormalities with clinical significance (frequency of occurrence, number of subjects experiencing the event).
To assess maximum observed plasma concentration (Cmax) following SAD and MAD doses | SAD phase - Day 1 at pre-dose, 0.25, 0.5, 1, 2, 4, 6, 8, 12, 15, 24, 36, 48, and 72 hours. MAD phase - Day 1 at pre-dose, 1, 2, 4, 6, 8, 12, and 24 hours after the first dose. Day 3 to Day 7 at pre-dose, 1, 2, 4, 6, 8, 12, and 24 hours.
  Cmax of FM101 in plasma will be calculated as applicable:
  SAD phase - cohort 1 to 6 , MAD phase - cohort 2
To assess area under plasma concentration-time curve from hour 0 to last sample following SAD and MAD doses | SAD phase - Day 1 at pre-dose, 0.25, 0.5, 1, 2, 4, 6, 8, 12, 15, 24, 36, 48, and 72 hours. MAD phase - Day 1 at pre-dose, 1, 2, 4, 6, 8, 12, and 24 hours after the first dose. Day 3 to Day 7 at pre-dose, 1, 2, 4, 6, 8, 12, and 24 hours.
  AUClast of FM101 in plasma will be calculated as applicable:
  SAD phase - cohort 1 to 6 , MAD phase - cohort 2
To assess area under plasma concentration-time curve from hour 0 to infinity following SAD and MAD doses | SAD phase - Day 1 at pre-dose, 0.25, 0.5, 1, 2, 4, 6, 8, 12, 15, 24, 36, 48, and 72 hours. MAD phase - Day 1 at pre-dose, 1, 2, 4, 6, 8, 12, and 24 hours after the first dose. Day 3 to Day 7 at pre-dose, 1, 2, 4, 6, 8, 12, and 24 hours.
  AUCinf of FM101 in plasma will be calculated as applicable:
  SAD phase - cohort 1 to 6 , MAD phase - cohort 2
To assess time to reach the maximum concentration in plasma (Tmax) following SAD and MAD doses | SAD phase - Day 1 at pre-dose, 0.25, 0.5, 1, 2, 4, 6, 8, 12, 15, 24, 36, 48, and 72 hours. MAD phase - Day 1 at pre-dose, 1, 2, 4, 6, 8, 12, and 24 hours after the first dose. Day 3 to Day 7 at pre-dose, 1, 2, 4, 6, 8, 12, and 24 hours.
  Tmax of FM101 in plasma will be calculated as applicable:
  SAD phase - cohort 1 to 6 , MAD phase - cohort 2
To assess terminal elimination rate constant (Kel) following SAD and MAD doses | SAD phase - Day 1 at pre-dose, 0.25, 0.5, 1, 2, 4, 6, 8, 12, 15, 24, 36, 48, and 72 hours. MAD phase - Day 1 at pre-dose, 1, 2, 4, 6, 8, 12, and 24 hours after the first dose. Day 3 to Day 7 at pre-dose, 1, 2, 4, 6, 8, 12, and 24 hours.
  Kel of FM101 in plasma will be calculated as applicable:
  SAD phase - cohort 1 to 6 , MAD phase - cohort 2
To assess terminal half-life (t1/2) following SAD and MAD doses | SAD phase - Day 1 at pre-dose, 0.25, 0.5, 1, 2, 4, 6, 8, 12, 15, 24, 36, 48, and 72 hours. MAD phase - Day 1 at pre-dose, 1, 2, 4, 6, 8, 12, and 24 hours after the first dose. Day 3 to Day 7 at pre-dose, 1, 2, 4, 6, 8, 12, and 24 hours.
  t1/2 of FM101 in plasma will be calculated as applicable: SAD phase - cohort 1 to 6 , MAD phase - cohort 2

SECONDARY OUTCOMES:
To evaluate the effect of food on the plasma Cmax of FM101 after a single dose | Day 1 pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 15, 24, 36, 48, and 72 hours post-dose.
  Cmax of FM101 under fasted and fed conditions will be calculated after a single dose.
To evaluate the effect of food on the plasma AUClast of FM101 after a single dose | Day 1 pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 15, 24, 36, 48, and 72 hours post-dose.
  AUClast of FM101 under fasted and fed conditions will be calculated after a single dose.
To evaluate the effect of food on the plasma AUCinf of FM101 after a single dose | Day 1 pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 15, 24, 36, 48, and 72 hours post-dose.
  AUCinf of FM101 under fasted and fed conditions will be calculated after a single dose.
To evaluate the effect of food on the plasma Tmax of FM101 after a single dose | Day 1 pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 15, 24, 36, 48, and 72 hours post-dose.
  Tmax of FM101 under fasted and fed conditions will be calculated after a single dose.
To evaluate the effect of food on the plasma Kel of FM101 after a single dose | Day 1 pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 15, 24, 36, 48, and 72 hours post-dose.
  Kel of FM101 under fasted and fed conditions will be calculated after a single dose.
To evaluate the effect of food on the plasma t1/2 of FM101 after a single dose | Day 1 pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 15, 24, 36, 48, and 72 hours post-dose.
  t1/2 of FM101 under fasted and fed conditions will be calculated after a single dose.

OTHER OUTCOMES:
Urine concentrations of FM101 in MAD cohort 2 | MAD phase - At pre-dose (within 12 hours prior to dosing), and over 0-6, 6-12, 12-18, and 18-24 hours post-dose collection intervals on Day 1 and Day 7.
  Cmax of FM101 in the urine will be calculated. MAD phase - cohort 2
Urine concentrations of M6, FM101's metabolite in MAD cohort 2 | MAD phase - At pre-dose (within 12 hours prior to dosing), and over 0-6, 6-12, 12-18, and 18-24 hours post-dose collection intervals on Day 1 and Day 7.
  Cmax of M6 in the urine will be calculated. MAD phase - cohort 2
Plasma concentrations of M6 in MAD cohort 2 | MAD phase - Day 1 at pre-dose, 1, 2, 4, 6, 8, 12, and 24 hours after the first dose. Day 3 to Day 7 at pre-dose, 1, 2, 4, 6, 8, 12, and 24 hours.
  Cmax of the plasma M6 will be calculated. MAD phase - cohor 2

CONTACTS AND LOCATIONS:
Overall Officials: WanSeok Jeong, MBA, Study Chair — Future Medicine Ltd.; Renger Tiessen, PhD, Principal Investigator — PRA Health Sciences
Locations (1):
- PRA health Sciences, Groningen, Gn, Netherlands

IPD SHARING:
Plan to Share IPD: No